CLINICAL TRIAL: NCT01709747
Title: A Phase 3, Open-Label, Single-Arm Study To Assess The Safety Of Hydromorphone Hydrochloride Delivered By Intrathecal Administration
Brief Title: Single-arm Study to Assess the Safety of Hydromorphone Hydrochloride by Intrathecal Administration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Piramal Critical Care, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS-HYD202US
Record Dates: First submitted 2012-09-04; First posted 2012-10-18 (Estimated); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Chronic Pain
Keywords: Hydromorphone Hydrochloride; Hydromorphone; Pain; Chronic Pain; Implantable Pump; Pump; Intrathecal
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Hydromorphone; Analgesics, Opioid; Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydromorphone Hydrochloride (Experimental): Hydromorphone hydrochloride for intrathecal administration, 12 months safety evaluation
  Interventions: Drug: Hydromorphone Hydrochloride; Device: Programmable Implantable pump

INTERVENTIONS:
Drug: Hydromorphone Hydrochloride — Opioid for chronic pain
  Other Names: Hydromorphone; Opioid
Device: Programmable Implantable pump — Device: Programmable Implantable pump
  Programmable Implantable pump delivering intrathecal hydromorphone

SUMMARY:
The purpose of this study is to evaluate the long-term safety of hydromorphone hydrochloride administered by intrathecal delivery.

DETAILED DESCRIPTION:
This is an open-label, single-arm safety study to evaluate the safety of hydromorphone hydrochloride given by continuous intrathecal infusion using an implantable pump device. This study will enroll both subjects on a current opioid intrathecal medication as well as naïve subjects now current on intrathecal opioid medications. All subjects currently on intrathecal opioid treatment will be converted from their current intrathecal therapy to intrathecal hydromorphone hydrochloride according to standard medical practice. After an optimal dose for pain relief is achieved, subjects will remain on therapy for a total of 12 months or until discontinuation from the study. During this continuous dosing period, dose adjustments (up or down) are permitted to manage pain or side effects provided a maximum dose of 10 mg/day is not exceeded. Subjects will be assessed for pain intensity using a visual analog scale of pain intensity (VASPI) instrument at each study visit.

Subjects will be evaluated for side effects and clinical complications associated with the use of intrathecal hydromorphone. Events will be classified by intrathecal drugs used and concentrations.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included:

1. Subjects must be at least 18 years of age and no more than 75 years old.
2. Clinically diagnosed with severe chronic pain for at least a 6-month period.
3. Subject is reasonably expected to benefit from intrathecal pain medication and has a programmable implantable intrathecal pump or meets clinical criteria for implantation of an intrathecal pump per Standard of Care.
4. Subject agrees to sign a Pain Treatment Agreement (Narcotic Contract) limiting narcotic prescriptions to the study medication prescribed by the investigator.
5. Subject must be cognitively intact and, in the opinion of the investigator, capable of participation in the trial.
6. Female subjects of child-bearing potential must agree to use a medically acceptable and effective double-barrier method of birth control.
7. Subjects who can receive an MRI if required by the study protocol.
8. Provides written Ethics Committee approved informed consent.
9. Willing to comply with all study procedures and requirements.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded:

1. Women who are pregnant or breast-feeding.
2. Subject has any known or suspected allergy to hydromorphone hydrochloride or to the materials of the infusion pump or intrathecal catheter.
3. Subject has a history of dependence and abuse of opioids, stimulants, alcohol, or benzodiazepines, as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria, within the past year (physical dependence on prescribed opioid analgesics is allowed but abuse of opioids according to DSM-IV is not permitted, i.e. opioid addiction for recreational use).
4. Subjects who show signs of active systemic infection.
5. Subjects with a metastatic cancer to the spinal canal or a known central nervous system contraindication to intrathecal therapy.
6. Subjects have a condition requiring diathermy procedures.
7. Subject has a life expectancy of less than 12 months.
8. Subjects who are unable or unwilling to return to all of the required follow-up visits.
9. As a result of medical review and physical examination, the Investigator considers the subject unfit for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rauck, MD, Principal Investigator — Carolinas Pain Institute
Locations (1):
- The Center for Clinical Research, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol states, "Approximately 350 subjects to be enrolled....... Additional subjects may be enrolled as deemed necessary to reach the study completion requirements for subjects on long term intrathecal hydromorphone hydrochloride therapy."
Groups:
- Hydromorphone Hydrochloride: Hydromorphone hydrochloride concentrations of 2mg/mL and 10 mg/mL for 0.1 mg/day to 10 mg/day based in dose titration, by intrathecal administration, 12 months safety evaluation
  Hydromorphone Hydrochloride: Opioid for chronic pain
  Programmable Implantable pump: Device: Programmable Implantable pump
  Programmable Implantable pump delivering intrathecal hydromorphone
Period: Overall Study
Arm/Group | Hydromorphone Hydrochloride
Started | 364
Completed | 287
Not Completed | 77

BASELINE CHARACTERISTICS:
Population: All Enrolled Subjects
Groups:
- Hydromorphone Hydrochloride: Hydromorphone hydrochloride 0.1 mg/day to 10 mg/day based in dose titration, by intrathecal administration, 12 months safety evaluation
  Hydromorphone Hydrochloride: Opioid for chronic pain
  Programmable Implantable pump: Device: Programmable Implantable pump
  Programmable Implantable pump delivering intrathecal hydromorphone
Arm/Group | Hydromorphone Hydrochloride
Number analyzed (Participants) | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220
  Male | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 356
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 4
  Black or African American | 16
  Native Hawaiian or Other Pacific Islander | 1
  White | 338
  Multi-racial (no primary race) | 2
  Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 364
Brief Pain Inventory (BPI) [Mean (Standard Deviation); unit: units on a scale] — Brief Pain Inventory (BPI): Pain Severity Measures, Scale: 0 = No Pain, 10 = Pain as bad as you can imagine; a high score indicates a worse outcome. Outcome is Mean Pain Severity score is calculated as the arithmetic mean of the Worst, Least, Average and Now severity scores. Population: Intent-to-Treat Population with non-missing data
  units on a scale
    number analyzed (Participants) | 358
    (all) | 5.44 (1.92)
Patient Global Impression of Change (PGIC) [Mean (Standard Deviation); unit: units on a scale] — Patient Global Impression of Change (PGIC): Scale: 7-point Likert scale, from 1 = No Change through 7 = A great deal better; a high score indicates a better outcome. Population: Intent-to-Treat (ITT) Population with non-missing values
  units on a scale
    number analyzed (Participants) | 357
    (all) | 4.24 (2.02)
Visual Analog Scale Pain Intensity (VASPI) [Mean (Standard Deviation); unit: mm] — Visual Analog Scale Pain Intensity (VASPI), Scale: 0 mm = No Pain, 100 mm = Unbearable Pain; high score is worse. Population: Intent-to-Treat (ITT) Population with non-missing assessment
  mm
    number analyzed (Participants) | 363
    (all) | 48.16 (26.69)

OUTCOME MEASURES:

1. Primary Outcome: Granulomas
Description: Subjects with Clinical Signs and Symptoms of Granuloma [Note: The primary endpoint of this trial is Safety. There is no formal efficacy assessment planned in this open-label safety study.]
Time Frame: 12 months
Population: All Enrolled Subjects
Measure: Count of Participants; unit: Participants
Groups:
- Hydromorphone Hydrochloride: Hydromorphone hydrochloride concentrations of 2 mg/mL and 10 mg/mL for 0.1 mg/day to 10 mg/day based in dose titration, by intrathecal administration, 12 months safety evaluation
  Hydromorphone Hydrochloride: Opioid for chronic pain
  Programmable Implantable pump: Device: Programmable Implantable pump
  Programmable Implantable pump delivering intrathecal hydromorphone
Arm/Group | Hydromorphone Hydrochloride
Number analyzed (Participants) | 364
Participants
  Subjects with Clinical Signs and Symptoms of Granuloma | 12
  Subjects without Clinical Signs and Symptoms of Granuloma | 352
  MRI Confirms Granuloma | 0
  Investigator Considers Signs and Symptoms to be Caused by Granuloma | 0

2. Secondary Outcome: Brief Pain Inventory (BPI) - Mean Pain Severity
Description: Change from Baseline in the Brief Pain Inventory (BPI). Pain Severity Measures, Scale: 0 = No Pain, 10 = Pain as bad as you can imagine; a high score indicates a worse outcome. Therefore, a negative change from baseline indicates a better outcome. Outcome is Mean Pain Severity score calculated as the arithmetic mean of the Worst, Least, Average and Now scores. A negative change indicates better outcome.
Time Frame: Early Termination/Final Visit through 12 months
Population: ITT (Intent to Treat) with non-missing Baseline and Early Termination/Final Visit assessment for computing change from baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydromorphone Hydrochloride
Number analyzed (Participants) | 334
units on a scale | -.20 (1.80)

3. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Change from Baseline in the Patient Global Impression of Change (PGIC). Scale: 7-point Likert scale, from 1 = No Change through 7 = A great deal better; a high score indicates a better outcome. Therefore, a positive change from baseline indicates a better outcome.
Time Frame: Early Termination/Final Visit through 12 months
Population: ITT (Intent to Treat) with non-missing Baseline and Final Visit assessment for computing change from baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydromorphone Hydrochloride
Number analyzed (Participants) | 337
units on a scale | 0.44 (2.13)

4. Secondary Outcome: Visual Analog Scale Pain Intensity (VASPI)
Description: Change from Baseline in Visual Analog Scale Pain Intensity (VASPI). Scale: 0 mm = No Pain, 100 mm = Unbearable Pain; high score is worse. Therefore, a negative change from baseline indicates a better outcome.
Time Frame: Early Termination/Final Visit through 12 months
Population: ITT (Intent to Treat) with non-missing Baseline and Final Visit assessment for computing change from baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Hydromorphone Hydrochloride
Number analyzed (Participants) | 344
mm | -0.41 (26.10)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Hydromorphone Hydrochloride
All-Cause Mortality (participants affected / at risk) | 7/364
Serious Adverse Events (participants affected / at risk) | 71/364
Other Adverse Events (participants affected / at risk) | 308/364
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydromorphone Hydrochloride (N=364)
Cellulitis (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 6
Sepsis (Infections and infestations) | 6
Pyelonephritis Acute (Infections and infestations) | 2
Bronchitis Viral (Infections and infestations) | 1
Gastroenteritis Viral (Infections and infestations) | 1
Implant Site Abscess (Infections and infestations) | 1
Implant Site Infection (Infections and infestations) | 1
Localised Infection (Infections and infestations) | 1
Necrotising Fasciitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia Bacterial (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Cardiac Failure Congestive (Cardiac disorders) | 3
Atrial Fibrillation (Cardiac disorders) | 2
Angina Unstable (Cardiac disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Cerebrospinal Fistula (Nervous system disorders) | 1
Cognitive Disorder (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Hepatic Encephalopathy (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Uraemic Encephalopathy (Nervous system disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis Ischaemic (Gastrointestinal disorders) | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Subdural Haematoma (Injury, poisoning and procedural complications) | 2
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Chest Pain (General disorders) | 2
Non-Cardiac Chest Pain (General disorders) | 2
Chronic Fatigue Syndrome (General disorders) | 1
Drug Withdrawal Syndrome (General disorders) | 1
Systemic Inflammatory Response Syndrome (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Mental Status Changes (Psychiatric disorders) | 3
Bipolar Disorder (Psychiatric disorders) | 1
Panic Attack (Psychiatric disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 3
Nephrolithiasis (Renal and urinary disorders) | 2
Cystitis Haemorrhagic (Renal and urinary disorders) | 1
Obstructive Uropathy (Renal and urinary disorders) | 1
Renal Colic (Renal and urinary disorders) | 1
Accelerated Hypertension (Vascular disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 1
Melas Syndrome (Congenital, familial and genetic disorders) | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Precancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hydromorphone Hydrochloride (N=364)
Back Pain (Musculoskeletal and connective tissue disorders) | 62
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 25
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 25
Urinary Tract Infection (Infections and infestations) | 25
Oedema Peripheral (General disorders) | 19
Pain (General disorders) | 19
Headache (Nervous system disorders) | 20
Nausea (Gastrointestinal disorders) | 51
Vomiting (Gastrointestinal disorders) | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT01709747/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/47/NCT01709747/SAP_001.pdf